CLINICAL TRIAL: NCT02992665
Title: Can Calcium Ionophore Application Enhance the ICSI Outcomes in Severe Male Factor Infertility?
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osama Saber Thabet Abdalmageed, Lecturer of OBGYN, Women Health Hospital, Assiut Univerisity, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CaII
Record Dates: First submitted 2016-12-11; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: In Vitro Fertilization; Male Factor Infertility
Keywords: Calcium ionophore; Fertilization; Sperm; Oocyte; ICSI

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ca ionophore (Experimental): Artificial activation of the oocytes using Calcium ionophore in the cases of severe male factor infertility.
  Interventions: Drug: Ca Ionophore A23187
- Placebo (Experimental): Placebo was used to control the group of Calcium ionophore
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ca Ionophore A23187 — Sibling oocytes are to be randomized to artificially activated using Calcium ionophore in cases with severely compromized semen parameters
  Other Names: Ca ionophore
  Arms: Ca ionophore
Other: Placebo — Placebo is used to control Ca ionophore group
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the impact of the use of calcium ionophore on the ICSI outcomes in couples with severe male factor infertility. Investigators conduct a randomized controlled trial on the sibling oocyte to justify the use of calcium ionophore in these cases.

DETAILED DESCRIPTION:
Elevation of calcium levels inside the oocyte is one of the most initial steps which takes place during normal fertilization (1). The interaction between the sperm and oocytes surface protein receptors may be the triggering event for oocyte activation during the process of fertilization (2). It is suggested that the process of intracellular Calcium elevation is triggered by binding of the sperm to the oocyte oolemma and hence the fertilization starts (3). Severe male factor couples might have compromised fertilization and pregnancy outcomes (4).

A prospective multicenter non-randomized study indicated that calcium ionophore could improve the fertilization as well as the clinical pregnancy rates in these patients (5). On the other hand, a randomized controlled trial did not find any significance for the use of calcium ionophore in the couples with poor ovarian reserve with regards the fertilization and clinical pregnancy rates (6). The purpose of this study is to determine the impact of the use of calcium ionophore on the ICSI outcomes in couples with severe male factor infertility. Investigators conduct a randomized controlled trial on the sibling oocyte to justify the use of calcium ionophore in these cases.

ELIGIBILITY:
Inclusion Criteria:

* Severe male factor infertility, Average response to COH,

Exclusion Criteria:

* Poor responders,

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Fertilization rate | 18 hours after injecting the sperms in the oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Osama Abdalmageed, Principal Investigator — Women health center, Assiut University
Locations (1):
- Osama Abdalmageed, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
According to the patient agreement.